CLINICAL TRIAL: NCT04421794
Title: Effects of One Electrical Strengthening Session on Foot Functions and Dynamic Postural Balance: a Randomised Controlled Trial in Single Blind
Brief Title: Effects of Foot Medial Arch Electrical Stimulation on Foot Functions and Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: La Tour Hospital (Other)
Responsible Party: Principal Investigator, Boris Gojanovic, Principal Investigator, La Tour Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020 - 00533
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Healthy
Keywords: Foot; Foot strength; Stability; Plantar pressure; Dynamic postural balance; Neuromuscular Electrical Stimulation; NMES; Transcutaneous Electrical Nerve Stimulation; TENS
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will be allocated to the intervention or control group using permuted block randomization with blocks of 4 or 6 patients on a 1:1 ratio.
Who Masked: Participant
Masking Description: This randomised controlled trial is in single blind. Participants will be informed about their treatment group after termination of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NMES group (Experimental): For the NMES group one portable stimulator (Compex 2, Medicompex SA, Ecublens, Switzerland) will deliver NEMS (15 min; 75 EMS contractions completed during the training session; rise time = 0.25 s and descending time = 0.75 s). In order to maximize muscle tension without accompanying detrimental effects on fatigue onset, biphasic symmetric regular-wave pulsed currents (85 Hz) lasting 400 μs will be delivered. Each 4-s steady tetanic stimulation will be followed by pause lasting 8-s, during which subjects will be submaximally stimulated at 4 Hz on the medial arch muscles. According to the recommendations, the two electrodes are placed behind the head of the first metatarsal to stimulate the medial arch intrinsic muscles. The goal is to attain the highest tolerable level of muscle contraction without discomfort during the 15 minutes and to provide a full tetanic contraction of the intrinsic foot muscles during the contraction time.
  Interventions: Device: NMES
- Control group (Placebo Comparator): For the control group the one portable stimulator (Compex 2, Medicompex SA, Ecublens, Switzerland) will be used to apply a stimulation of 15 minutes considered by TENS at the lowest intensity detectable by the participant in order to not influence the outcomes of interest. Our aim is to strengthen IFM which is not the role of TENS. The two electrodes will be placed on the dominant foot, at the same place than those for the NMES group.
  Interventions: Device: TENS

INTERVENTIONS:
Device: NMES — Neuromuscular Electrical Stimulation (NMES) is a non pharmacological intervention that sends electrical impulses to nerves leading to muscle contraction. The electrical stimulation can increase strength and is often used to re-educate or re-train muscles.
  Arms: NMES group
Device: TENS — Transcutaneous electrical nerve stimulation (TENS) is a nonpharmacological intervention that activates a complex neuronal network to reduce pain by activating descending inhibitory systems in the central nervous system to reduce hyperalgesia.
  Arms: Control group

SUMMARY:
The aim of this study is to investigate the immediate effects of sole session of foot medial arch' NMES on foot strength, arch stability, static plantar pressure distribution and dynamic postural balance.

DETAILED DESCRIPTION:
The study design is a randomised controlled trial in population with pronated feet. The aim of this study is to investigate the immediate effects of sole session of foot medial arch' NMES on foot strength, arch stability, static plantar pressure distribution and dynamic postural balance. This is the 2nd study to investigate the effect one session as previous study showed immediate effect on plantar pressure distribution on the midfoot and durable effect at 2 months follow-up. However, no studies investigated the effects on others parameters than plantar pressure.The general objective of our study is to question electrical stimulation as a modality for foot strengthening to enhance dynamic postural balance and foot functions.

ELIGIBILITY:
Inclusion Criteria:

* Foot Posture Index (FPI) between +6 à +12 (slight pronation / increased pronation)

Exclusion Criteria:

* History of ankle or foot sprain or pain within the last 3 months
* Fracture in the leg or in the foot that occurred during the last year
* Severe foot deformity
* Self-reported disability due to neuromuscular impairment in the lower extremity
* Neurological or vestibular impairment that affected balance (diabetes mellitus, lumbosacral radiculopathy, a soft tissue disorder such as Marfan or Ehlers-Danlos syndrome)
* Any absolute contraindication to NMES (pacemaker, seizure disorders, pregnancy)
* Experience of NMES at the foot region or foot core strengthening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Foot strength | Before and immediately after intervention
  The change of foot strength that will be measured on a pressure platform on the dominant foot before and after intervention (NMES or TENS). This primary outcome will be also measured on the non-dominant foot to assess cross effects.

SECONDARY OUTCOMES:
Dynamic postural balance | Before and immediately after intervention
  The secondary outcomes include the change of dynamic postural balance in the posterior direction on the dominant foot. All measurements will be performed on the non-dominant foot to assess cross effects. To assess dynamic postural balance performance, we will use the Star Excursion Balance Test (SEBT). The star excursion balance test (SEBT) is a measure of dynamic balance with good to excellent test-retest reliability. The test will be conducted in the anterior, posterior-lateral and posterior-medial directions. The SEBT will be performed with the subject standing barefoot so that the distal end of the longest toe of the stance foot will be placed at the center of the grid. They will have to maintain a single-leg stance while reaching with the contralateral leg to touch as far as possible along the direction by a light touch. The reached distances will be normalized to the respective stance-limb length (anterior superior iliac spine to the inferior border of the medial malleolus).
Arch stability | Before and immediately after intervention
  The secondary outcomes include the change of arch stability on the dominant foot. This measurement will be performed on the non-dominant foot to assess cross effects. The sit-to-stand double-leg navicular drop test will be used to evaluate longitudinal arch stability. Participants will sit on a chair with their hips, knees, and ankles bent to 90° and the feet resting on the floor. The inferior border of the prominent tuberosity of the navicular bone will be palpated and marked with a pen. Next, the distance of the marked navicular point to the ground in a seated position will be measured using a steel ruler (resolution: 0.5 mm). Then, we will ask the subject to stand barefoot on a 4-in (10.16-cm) box, placing all weight on the foot being measured, while the other foot rested lightly on the box. Finally, the difference between the two measures (sitting - standing) will be calculated and defined as navicular drop (ND).
Static plantar pressure distribution | Before and immediately after intervention
  The secondary outcomes include the change of arch stability on the dominant foot. In this study the evaluation of the longitudinal arch of the foot will be made with the use of the Zebris FDM-S dynamometric platform. It will describe foot arch assessment based on the AI calculated on the basis of discretized measurements of distribution of forces on the ground, by means of the platform.
  According to this theory, a static arch pressure index (SAPI) will be measured by utilizing the average/maximal foot pressure distribution during static single leg standing of 30 seconds with their arms along the body while the subject will have one foot on a Zebris platform. Based on distribution of pressure on the entire foot the SAPI will be calculate as the ratio of the midfoot pressure distribution relative to the whole foot pressure distribution excluding the toes.

CONTACTS AND LOCATIONS:
Overall Officials: Boris Gojanovic, MD, Principal Investigator — La Tour Hospital
Locations (1):
- La Tour Hospital, Meyrin, Switzerland

IPD SHARING:
Plan to Share IPD: No